CLINICAL TRIAL: NCT02303392
Title: A Dose Escalation Study of Selinexor (KPT-330), a Selective Inhibitor of Nuclear Export, and Ibrutinib, a Bruton's Tyrosine Kinase Inhibitor, in Patients With Relapsed and Refractory Chronic Lymphocytic Leukemia or Aggressive Non-Hodgkin Lymphoma
Brief Title: Selinexor and Ibrutinib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Aggressive Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer Woyach (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Woyach, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14087; NCI-2014-01493 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — selinexor; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selinexor, ibrutinib) (Experimental): Patients receive ibrutinib PO on days 8-28 of course 1 and on days 1-28 on subsequent courses and selinexor PO BID weekly on day 1 or bi-weekly on days 1 and 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selinexor; Drug: Ibrutinib; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of selinexor when given together with ibrutinib in treating patients with chronic lymphocytic leukemia or aggressive non-Hodgkin lymphoma that has returned after a period of improvement or does not respond to treatment. Drugs used in chemotherapy, such as selinexor, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving selinexor together with ibrutinib may be a better treatment for chronic lymphocytic leukemia or aggressive non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose for the combination of selinexor and ibrutinib in patients with relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia(SLL)/B-cell prolymphocytic leukemia (PLL) or aggressive non-Hodgkin lymphoma (NHL).

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of the combination of selinexor and ibrutinib in patients with relapsed or refractory CLL/SLL/PLL or aggressive NHL.

II. To characterize the pharmacokinetic (PK) properties of the combination of selinexor and ibrutinib in patients with relapsed or refractory CLL/SLL/PLL or aggressive NHL.

III. To obtain preliminary evidence on efficacy of the combination of selinexor and ibrutinib in patients with relapsed or refractory CLL/SLL/PLL or aggressive NHL.

IV. To obtain preliminary evidence of response in CLL/SLL/PLL and diffuse large B-cell lymphoma (DLBCL) patients receiving the combination of selinexor and ibrutinib as related to CLL/SLL/PLL karyotype and immunoglobulin variable heavy chain (IgVH) mutational status and DLBCL subtype, respectively.

V. To evaluate the inhibition of the B-cell receptor signaling pathway in patients with relapsed or refractory CLL/SLL/PLL who receive the combination of selinexor and ibrutinib.

VI. To evaluate the change in localization of tumor suppressor and growth regulation proteins in patients with relapsed or refractory CLL/SLL/PLL following treatment with selinexor in general and as related to response.

VII. To preliminarily assess potential causes for primary and secondary resistance to selinexor and ibrutinib.

VIII. To measure intracellular levels of selinexor and metabolites in peripheral blood mononuclear cells and to identify how this relates to pharmacodynamics effects and clinical outcomes.

OUTLINE: This is a dose-escalation study of selinexor.

Patients receive ibrutinib orally (PO) on days 8-28 of course 1 and on days 1-28 on subsequent courses and selinexor PO twice daily (BID) weekly on day 1 or bi-weekly on days 1 and 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* A histologically confirmed diagnosis of CLL according the International Workshop on CLL/SLL/B-cell PLL or variant of these (IWCLL or World Health Organization [WHO] Criteria) and meet criteria for treatment or have need for cytoreduction for stem cell transplantation or alternative cell therapy; OR
* A histologically confirmed diagnosis of mantle cell lymphoma (MCL) or diffuse large B-cell lymphoma (DLBCL) de novo or in the setting of transformation from an indolent lymphoma (including DLBCL not otherwise specified) according to the World Health Organization criteria for diagnosis of NHL; AND
* Patients must have received at least one prior therapy for CLL or NHL, need additional treatment, and meet criteria for relapsed or refractory disease; they may not be a candidate for curative therapy; relapsed disease is defined as a patient who previously achieved a complete remission (CR) or a partial remission (PR), but after a period of six or more months demonstrates evidence of disease progression; refractory disease is defined as progression within six months of the last anti-leukemic or anti-lymphoma therapy, or any response less than a CR or PR
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients with NHL must have objective, documented evidence of disease prior to study entry
* Platelet count >= 50,000/mm^3 in the absence of bone marrow involvement; patients with bone marrow involvement only require a platelet count of 30,000/mm^3
* Absolute neutrophil count >= 1000/mm^3 in the absence of bone marrow involvement
* Creatinine clearance (as calculated by Cockroft Gault equation = [140-age] * mass [kg]/[72 * creatinine mg/dL) >= 30mL/min
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 times upper limit of normal (ULN)
* Total bilirubin =< 2.0 x ULN
* Female patients capable of reproduction and male patients who have partners capable of reproduction must agree to use an effective contraceptive method during the course of the study and for 2 months following the completion of their last treatment
* Female of childbearing potential must have a negative serum beta-human chorionic gonadotropin (HCG) pregnancy test result within 3 days of first study dose; female patients who are surgically sterilized or who are > 45 years old and have not experienced menses for > 2 years may have beta-HCG pregnancy test waived
* Patients who are hepatitis B polymerase chain reaction (PCR) negative who have a recent (< 6 month) history of intravenous immunoglobulin (IVIG) therapy are eligible; patients with a history of hepatitis B (surface antigen or core antibody positive and PCR positive) must take lamivudine or equivalent drug during study therapy and for one year after completion of all therapy; patients on IVIG who are core antibody positive but PCR negative are not mandated to take prophylaxis
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are concurrently receiving any other investigational agents
* Patients who have received:

  * Radiation or chemotherapy =< 4 weeks
  * Mitomycin C, nitrosureas, or radio-immunotherapy =< 6 weeks, or
  * Immunotherapy or targeted therapy (such as kinase inhibitors) =< 2 weeks prior to cycle 1 day 1(except patients already on ibrutinib)
  * Palliative steroids for disease related symptoms are allowed as long as dose is tapered down to an equivalent of =< 10 mg of oral prednisone daily on cycle 1 day 1
* Patients who have underwent autologous or allogeneic stem cell transplant =< 4 weeks prior to cycle 1 day 1 or have active graft-versus-host disease are excluded
* Patients unable to swallow capsules, those with uncontrolled vomiting or diarrhea or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as: malabsorption syndrome, resection of the small bowel, or poorly controlled inflammatory bowel disease affecting the small intestine
* Patients who are 20% below their ideal body weight
* Patients must not be receiving systemic anticoagulation with warfarin; patients must be off warfarin for 30 days prior to enrollment; patients who require anticoagulation with an agent other than warfarin will not be excluded, but must be reviewed by the principal investigator prior to enrollment
* As ibrutinib is extensively metabolized by cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5), and patients must not require continued therapy with a strong inhibitor or inducer of CYP3A4/5
* Patients with active human immunodeficiency virus (HIV) or hepatitis B or C
* Patients with secondary malignancy that requires active systemic therapy that will interfere with interpretation of efficacy or toxicity of selinexor; (Note: patients with basal or squamous skin carcinoma, cervical carcinoma in situ, localized breast cancer requiring hormonal therapy or localized prostate cancer (Gleason score < 5 are allowed)
* Patients with active known central nervous system (CNS) involvement of CLL or lymphoma; (patients with history of CNS CLL or lymphoma now in remission are eligible for the trial)
* Patients who are pregnant or breast feeding; breastfeeding should be discontinued if the mother is treated with selinexor
* Patients must have recovered all toxicities from prior therapy or radiation to grade 1 or less (excluding alopecia)
* Patients may not have had major surgery within 10 days of enrollment, or minor surgery within 7 days of enrollment; examples of minor surgery include dental surgery, insertion of a venous access device, skin biopsy, or aspiration of a joint; the decision about whether a surgery is major or minor can be made at the discretion of the treating physician
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with markedly decreased visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Woyach, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephens DM, Huang Y, Ruppert AS, Walker JS, Canfield D, Cempre CB, Fu Q, Baker S, Hu B, Shah H, Vadeboncoeur R, Rogers KA, Bhat S, Jaglowski SM, Lockman H, Lapalombella R, Byrd JC, Woyach JA. Selinexor Combined with Ibrutinib Demonstrates Tolerability and Safety in Advanced B-Cell Malignancies: A Phase I Study. Clin Cancer Res. 2022 Aug 2;28(15):3242-3247. doi: 10.1158/1078-0432.CCR-21-3867. PMID 35608822
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 2015 until July 2019
Pre-assignment Details: Patients with diagnoses with chronic lymphocytic leukemia (CLL) or non-Hodgkin Lymphoma (NHL) (the NHL arm comprises of diagnoses of Richter transformation (RT), diffuse B-cell lymphoma (DBCL), and mantle cell lymphoma (MCL)) were enrolled
Groups:
- Chronic Lymphocytic Leukemia (CLL): Patients receive ibrutinib PO on days 8-28 of course 1 and on days 1-28 on subsequent courses and selinexor PO BID weekly on day 1 or bi-weekly on days 1 and 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Selinexor: Given PO
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
- Non-Hodgkin Lymphoma (NHL): Patients receive ibrutinib PO on days 8-28 of course 1 and on days 1-28 on subsequent courses and selinexor PO BID weekly on day 1 or bi-weekly on days 1 and 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Selinexor: Given PO
  Ibrutinib: Given PO
Period: Overall Study
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL) | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 17
  >=65 years | 5 | 12 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34
Number of prior therapies [Count of Participants; unit: Participants]
  1 | 3 | 2 | 5
  2 | 2 | 1 | 3
  3-8 | 11 | 10 | 21
  10-14 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose for Selinexor
Description: To determine the maximum tolerated dose for the combination of selinexor and ibrutinib in patients with relapsed or refractory chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia(SLL)/B-cell prolymphocytic leukemia (PLL) or aggressive non-Hodgkin lymphoma (NHL).
Time Frame: Day 28
Measure: Number; unit: mg
Arm/Group | Treatment (Selinexor, Ibrutinib)
Number analyzed (Participants) | 34
mg | 40

2. Secondary Outcome: Number of Participants With Toxicities Graded by CTCAE V4 That Are Grade 3 or Higher
Description: Toxicities will be tabulated by type and grade and displayed in summary form. In addition, the number of courses started/completed, number of patients requiring dose reductions, and the reason for going off treatment may be summarized to assess treatment tolerability.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Groups:
- Non-Hodgkin Lymphoma (NHL): Patients receive ibrutinib PO on days 8-28 of course 1 and on days 1-28 on subsequent courses and selinexor PO BID weekly on day 1 or bi-weekly on days 1 and 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Selinexor: Given PO
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
Number analyzed (Participants) | 16 | 18
Participants
  Thrombocytopenia | 6 | 2
  Anemia | 2 | 4
  Neutropenia | 4 | 1
  Lymphocyte count increased | 3 | 1
  Lymphopenia | 1 | 6
  Nausea | 1 | 0
  Diarrhea | 1 | 1
  Hypertension | 5 | 4
  Joint/Bone Pain | 1 | 0
  Hyponatremia | 3 | 2
  Pneumonia | 1 | 2
  Hyperglycemia | 1 | 1
  Fall | 2 | 0
  Cataract | 1 | 1
  Cognitive Disturbance | 1 | 0
  Hypophosphatemia | 1 | 2
  Death | 1 | 2
  Hypoxia | 0 | 2

3. Secondary Outcome: Clinical Response Defined as Those With CR or PR
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of patients
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
Number analyzed (Participants) | 16 | 18
percentage of patients | 44 | 22

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS): PFS calculated from the date of study enrollment to disease progression or death, whichever occurs first. Patients who do not progress or die will be censored at the time of last contact with response assessment by physical exam and laboratory studies.
Time Frame: Date of study enrollment to disease progression or death, whichever occurs first assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
Number analyzed (Participants) | 16 | 18
months | 8.9 [3.9 to 16.1] | 2.7 [0.7 to 5.4]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) calculated from the date of study enrollment to death. Patients who do not die will be censored at the time of last contact. This will be analyzed in each cohort independently
Time Frame: Date of study enrollment to death assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
Number analyzed (Participants) | 16 | 18
months | 58.9 [19.6 to 58.9] | 5.1 [3.0 to 14.8]

6. Primary Outcome: Maximum Tolerated Dose for Ibrutinib
Description: as for outcome 1
Time Frame: Day 28
Measure: Number; unit: mg
Arm/Group | Treatment (Selinexor, Ibrutinib)
Number analyzed (Participants) | 34
mg | 420

ADVERSE EVENTS:
Time Frame: All patients must be carefully monitored for AEs, including clinical laboratory tests. AEs should be assessed in terms of their seriousness, intensity, and relationship to the study drug. For consistency, events are to be graded using the CTCAE version 4.0 from start of study to completion for up to 4 years.
Description: CTCAE version 4.0 is used to grade all adverse events and to provide management guidelines for administrational toxicity. Adverse events from all arms are reported together as participants on all arms received the same treatment regimen.
Arm/Group | Chronic Lymphocytic Leukemia (CLL) | Non-Hodgkin Lymphoma (NHL)
All-Cause Mortality (participants affected / at risk) | 1/16 | 4/18
Serious Adverse Events (participants affected / at risk) | 6/16 | 7/18
Other Adverse Events (participants affected / at risk) | 16/16 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia (CLL) (N=16) | Non-Hodgkin Lymphoma (NHL) (N=18)
Colonic Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 1 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Death, NOS (General disorders) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Infections and Infestations-other (Infections and infestations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (3)
Multi-organ Failure (General disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders, Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
E. coli bacteremia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Lymphocytic Leukemia (CLL) (N=16) | Non-Hodgkin Lymphoma (NHL) (N=18)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 3 (3)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (8) | 7 (13)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Alkaline Phosphatase increased (Investigations) | 5 (10) | 4 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (9) | 1 (1)
Altered Mental Status (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 14 (39) | 14 (48)
Anorexia (Metabolism and nutrition disorders) | 8 (11) | 10 (12)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (7) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Atrial Flutter (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Autoimmune disorder (Sjogren's syndrome) (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Benign Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Prostatic Hypertrophy (BPH) (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Blood Blisters (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Blurry Vision (Eye disorders) | 4 (6) | 4 (4)
Bone spur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Brain fog (Nervous system disorders) | 1 (1) | 0 (0)
Brittle nails (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 6 (8) | 8 (9)
Bruxism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac disorder - other Chest Pressure, intermittent (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (4) | 5 (5)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Chest heaviness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest Tightness (Cardiac disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Chills (Intermittent) (General disorders) | 1 (1) | 0 (0)
Chronic Fatigue (General disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 1 (1) | 0 (0)
Cold sore (Infections and infestations) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (8) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 7 (8)
Creatinine Increased (Investigations) | 6 (15) | 4 (9)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (4)
Diabetes Mellitus (Endocrine disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (16) | 10 (16)
Dizziness (Nervous system disorders) | 4 (5) | 4 (4)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (6) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 7 (9)
Early satiety (Gastrointestinal disorders) | 1 (1) | 1 (1)
Edema (General disorders) | 3 (3) | 4 (4)
Enlarged Left Lingual Tonsil (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Eustachian Tube Dysfunction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Eye disorders, other - itching, without redness, swelling, or watering (Eye disorders) | 1 (1) | 0 (0)
Eye Infection (Eye disorders) | 1 (3) | 2 (2)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fatigue (General disorders) | 13 (26) | 13 (24)
Fever (General disorders) | 4 (5) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu Like Symptoms (General disorders) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (3)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 8 (8) | 3 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clay colored stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ground Glass Opacities (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (16) | 3 (6)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (17) | 5 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (9) | 5 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypertension (Vascular disorders) | 12 (31) | 15 (32)
Hyperuricemia (Metabolism and nutrition disorders) | 8 (11) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9) | 7 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (17) | 3 (4)
Hypogonadism (Endocrine disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 4 (15) | 7 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hypoproteinemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Increased BNP (Cardiac disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (4) | 0 (0)
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
International normalized ratio (INR) increased (Investigations) | 1 (1) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8) | 3 (4)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Intermittent Ocular Migraine (Eye disorders) | 1 (2) | 0 (0)
Intermittent Oral Sores (Infections and infestations) | 1 (1) | 0 (0)
Intermittent Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Iron deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Knee injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Knee sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lactate Dehydrogenase (LDH) increased (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Left index finger knuckle purple discoloration with a scab, secondary to trauma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Localized edema (General disorders) | 2 (2) | 6 (8)
Low Vitamin D (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lower Lip Lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 3 (5) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Lymphocyte count increased (Investigations) | 11 (14) | 4 (7)
Lymphocyte count decreased (Investigations) | 2 (12) | 10 (29)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 5 (6) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Nail splitting (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (2)
Nausea (Gastrointestinal disorders) | 11 (19) | 11 (18)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (24) | 7 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 6 (7)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 3 (4) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 7 (8) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Platelet count decreased (Investigations) | 15 (48) | 13 (30)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Prostate Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Pulsatile Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Restless Leg Symptoms (Nervous system disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right small finger knuckle purple discoloration with a scab, secondary to trauma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shin cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 6 (7) | 5 (7)
Bug bite hypersensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Infection (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Skin splitting on fingertips (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Subconjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Superficial Venous Thrombus (Left Radial Vein) (Vascular disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 6 (10) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 4 (4) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 3 (5)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Visual aura (Eye disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (8) | 5 (6)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Weight gain (Investigations) | 2 (5) | 1 (4)
Weight loss (Investigations) | 5 (9) | 5 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 5 (13) | 9 (13)
Allergic Reaction (Immune system disorders) | 0 (0) | 2 (2)
Anterior uveitis (Eye disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's Esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
C. difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chronic Sciatic Nerve Pain (Nervous system disorders) | 0 (0) | 1 (1)
Colon Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Resection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intermittent Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
DLBCL (richter's transformation) (General disorders) | 0 (0) | 1 (1)
Dyslipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Eye disorder - other, decreased visual acuity right eye (Eye disorders) | 0 (0) | 1 (1)
Facial nerve disorder (cranial nerve VII dysfunction) (Nervous system disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Fluid build up in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypogammaglobulinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular Pucker (Eye disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
MSSA Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Muscle weakness in lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
palpable lymph node (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Prothrombin time prolonged (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Red spots on arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal disorder, other (Renal and urinary disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Right Eye Swelling (Eye disorders) | 0 (0) | 1 (1)
Right vision changes (Eye disorders) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Skin graft (leg to arm & chest) (Surgical and medical procedures) | 0 (0) | 1 (1)
Intermittent skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Split Fingertips and Toes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sudden onset of slurred speech and difficulty with word forming (intermittent) (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent Sweats (General disorders) | 0 (0) | 1 (1)
Thrush in the mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Total Knee Arthroplasty (Right) (Surgical and medical procedures) | 0 (0) | 1 (2)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tubular Adenoma of the Colon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract obstruction - with bilateral hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Vascular Disorder, Other - diffuse Petechia (Vascular disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02303392/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT02303392/ICF_001.pdf